CLINICAL TRIAL: NCT02961530
Title: Effect of Rehabilitation Programs Based on Eccentric Exercise of Knee Extensor Muscles in Isotonic and Isokinetic Conditions After Partial Menisectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Marlon Francys Vidmar, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUHSPortoAlegre_IV
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Meniscal Tear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1. (Experimental): The participants randomly allocated to this arm will undergo a muscular rehabilitation program based on the isokinetic eccentric exercise for the extensor muscles of the operated knee.
  The contralateral non-operated lower limb will be used as control, so it will not undergo any muscular rehabilitation program.
  Interventions: Other: Isokinetic eccentric exercises
- Group 2. (Active Comparator): The participants randomly allocated to this arm will undergo a muscular rehabilitation program based on the isotonic eccentric exercise for the extensor muscles of the operated knee.
  The contralateral non-operated lower limb will be used as control, so it will not undergo any muscular rehabilitation program.
  Interventions: Other: Isotonic eccentric exercises

INTERVENTIONS:
Other: Isokinetic eccentric exercises — The individuals of both groups will be submitted to the same physiotherapeutic protocol with objectives of analgesia, reduction of edema, recovery of range of motion, proprioception and functionality.
  15 days after partial menisectomy, subjects randomly allocated to this arm will be submitted to a muscle rehabilitation program based on isokinetic eccentric exercise lasting six weeks, with training frequency of two sessions per week, separated by a minimum interval of 72 hours.
  Arms: Group 1.
Other: Isotonic eccentric exercises — The individuals of both groups will be submitted to the same physiotherapeutic protocol with objectives of analgesia, reduction of edema, recovery of range of motion, proprioception and functionality.
  15 days after partial menisectomy, subjects randomly allocated to this arm will be submitted to a muscle rehabilitation program based on isotonic eccentric exercise lasting six weeks, with training frequency of two sessions per week, separated by a minimum interval of 72 hours.
  Arms: Group 2.

SUMMARY:
A randomized clinical trial involving 32 individuals submitted to partial menisectomy will be conducted.

Participants will be randomized into: Group I, submitted to a muscular rehabilitation program based on eccentric isokinetic exercise; and Group II, submitted to a muscular rehabilitation program based on eccentric isotonic exercise. Concomitantly with the muscular rehabilitation protocols, individuals will undergo the same physiotherapeutic protocol with analgesia, edema reduction, range of motion, proprioception and functionality goals. Muscle rehabilitation programs based on eccentric isotonic and isokinetic exercise will begin 15 days after partial menisectomy. The programs will last six weeks, with training frequency of two sessions per week, separated by a minimum interval of 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged between 18 and 40 years;
* Recreational athletes;
* Unilateral partial meniscal tear;
* Partial meniscectomy by video-arthroscopy within 90 days after injury;
* Male subjects;
* Classification of body mass index up to pre-obese (25.0 - 29.9 kg / m2);
* Not undergoing any strength training program for the lower limbs in the six months prior to the study;
* Acceptance of individuals in participating in the procedures proposed by the research.

Exclusion Criteria:

Repeated meniscal tear; Associated ligament injuries; Previous history (<6 months) of musculoskeletal lesions in the thigh; Patellar tendinopathy; Patellofemoral pain syndrome; Respiratory or cardiovascular conditions that limit the performance of exercises; Users of dietary supplements or anabolic steroids

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The femoral quadriceps muscle mass through nuclear magnetic resonance imaging | Change from baseline and six weeks after intervention protocol

SECONDARY OUTCOMES:
Performance of knee extensors through computerized dynamometry | Change from baseline and six weeks after intervention protocol
Functionality of the individuals through Lysholm score | Change from baseline and six weeks after intervention protocol
Functionality of the individuals through single and triple hop test | Change from baseline and six weeks after intervention protocol

CONTACTS AND LOCATIONS:
Overall Officials: Marlon F Vidmar, MSc, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil